CLINICAL TRIAL: NCT07355803
Title: EVA-study on Catheter Selection Criteria at Start of Self-catheterization
Brief Title: Define Final Selection Choice Criteria for a Coloplast Catheter Ensuring Highest Patient Satisfaction Via Surveys (EVA).
Acronym: EVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast NV/SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVA-Belgium
Record Dates: First submitted 2025-12-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Bladder Disorder; Non-Neurogenic Bladder; Bladder Dysfunction; Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coloplast (Experimental): The study population will consist of adults with neurogenic and non-neurogenic bladder issues, newly initiated at ISC, and users of Coloplast catheters.
  The subject's participation in the study does not involve any additional examinations compared to the usual management of a patient. Only study questionnaires are used.
  Patients are free to make the decision to change catheters during follow-up if the initially chosen catheter is not suitable for them. In this case, this change will be documented as well as the model and brand of the new catheter chosen, and the patient will continue the study normally.
  Interventions: Other: Questionnaires : Patient questionnaire on catheter use and satisfaction, IC-Di-Q, and I-CAT

INTERVENTIONS:
Other: Questionnaires : Patient questionnaire on catheter use and satisfaction, IC-Di-Q, and I-CAT — The study will be conducted in three visits (inclusion visit (V1), visit between 3 and 12 weeks (V2), visit at 6 months (V3)) during which investigators will collect data specific to the self-catheterization methods and to the use of catheters from the SpeediCath range or the Luja catheters, as well as a set of patient questionnaires. In the case of a catheter change during follow-up, the model and brand of the new catheter will be documented, and the participant will continue the study.

SUMMARY:
Understanding the Coloplast Intermittent Catheter Selection Study:

This study aims to understand how adults who need to use catheters to empty their bladder by themselves decide which Coloplast catheter works best for them. The two types of catheters studied are called SpeediCath and Luja.

Why is this study being done? The study wants to find out which catheter type helps people feel most satisfied when they start to use it on their own. It also looks at why people choose their catheter at the beginning, how happy they are with it over the first six months, and what problems they might face using it.

Who can join the study?

* Adults aged 18 or older who have bladder problems and need to empty their bladder using a catheter.
* People who have been trained on how to use a catheter.
* People who have chosen to use either SpeediCath or Luja catheters from Coloplast.
* People who can perform the catheterization themselves at least two times per day.

Certain people cannot join, such as pregnant women, anyone who cannot give consent, or those who have trouble filling out questionnaires.

What will happen in the study?

Participants will visit the study center three times:

* At the start (to select their catheter and answer questions about the reasons for the specific catheter selection)
* After 3 to 12 weeks (to share their perception on the impact of the used catheter)
* After 6 months (to measure final satisfaction and any difficulties)

If a participant changes to a different catheter type or catheter brand during the study, this will be recorded, and they will continue in the study.

How will this study help? The information gathered will help healthcare providers understand what matters most to people when selecting a catheter. This can improve how catheters are recommended and support patients better during self-catheterization and improve treatment adherence and compliance.

DETAILED DESCRIPTION:
This multicentre prospective study examines the detailed clinical and technical aspects of intermittent self-catheterisation (ISC) training and catheter selection among adults with neurogenic or non-neurogenic bladder dysfunctions, such as those caused by spinal cord injuries, multiple sclerosis, Parkinson's disease, stroke, or pelvic surgeries.

Medical rationale :

ISC is the standard method for managing bladder emptying disorders, particularly in cases of urinary retention or incomplete voiding due to subvesical obstruction, aiming to reduce morbidity from vesico-sphincter dysfunctions and enhance patient independence. Training typically occurs during hospital admission by nursing staff or specialists, followed by outpatient monitoring at 3-12 weeks and 6 months to assess technique mastery, catheter suitability, compliance (frequency, volume), and complications. Despite expert training, long-term adherence remains challenging due to psychological barriers and equipment mismatches, underscoring the need for patient-involved catheter selection.

Technical catheter details :

Coloplast's SpeediCath® range includes hydrophilic, ready-to-use catheters differentiated by length, flexibility, shape, and ergonomics: Standard (40 cm men/20 cm women), Compact (no-touch for discretion), Compact Eve (triangular female design), Flex (multi-directional tip for men), with some available as pre-connected sets. Newer Luja™ catheters incorporate Micro-hole Zone Technology (>80 micro-holes in men, >50 in women) to minimise flow-stops, residual urine, and urinary tract infection (UTI) risk-addressing common issues where conventional eyelet catheters cause mucosa adhesion and incomplete emptying. Evidence shows hydrophilic catheters reduce urethral trauma and improve quality of life, with SpeediCath® demonstrating faster, more discreet use versus non-ready-to-use alternatives, and Luja/MHZC outperforming comparators in flow dynamics and user ratings. All are Class I sterile CE-marked devices manufactured by Coloplast A/S.

Study design and data collection This descriptive interventional cohort embeds questionnaire-based assessments into routine care across ~7 sites (urology/rehabilitation centres), targeting 107 patients for 6-month follow-up after a 6-month inclusion period. Beyond basic selection criteria, data capture socio-demographics (age, living status, education, occupation), clinical factors (pathology severity, USP symptom scores, anorectal dysfunction, meatus accessibility, urethral sensitivity, concomitant treatments), and ISC specifics (training location/duration, prescription frequency, solo vs. combined with micturition).

Validated tools include I-CAT (14 items, score 0-56 for ISC acceptance) and IC-Di-Q (13 items on pain, blockage, bleeding, spasticity frequency/intensity); a custom questionnaire details choice drivers (e.g., ease, discretion, nurse advice). Statistical plans use SAS V9.4 for descriptive stats, logistic regressions identifying predictors of final choice/adherence, with per-protocol exclusions for major deviations and precision ±4.25-9.5% for key frequencies. No blinding applies to this open-label routine care evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged eighteen years or older;
* Written informed consent;
* Subject affiliated with a social security scheme or beneficiary;
* Subject with neurogenic or non-neurogenic bladder issues, justifying the implementation of intermittent self-catheterisation (ISC) to clean out the bladder;
* Subject who received his/her initial ISC training at the time of inclusion;
* Subject for whom the expected ISC duration is at least six months;
* Subject for whom at least two types of Coloplast catheters have been introduced and who has chosen to use Coloplast catheters as the first catheter for self-catheterisation;
* Subject able to independently conduct ISC;
* Subject for whom the healthcare professional has recommended to conduct ISC at least four times per day.

Exclusion Criteria:

* Vulnerable subject with regard to the current regulation:

  * Pregnant, parturient or breast-feeding woman;
  * Subject deprived of freedom by judicial, medical or administrative decision;
  * Underage subject;
  * Subject is legally protected or unable to express his/her consent;
  * Subject not affiliated with or not a beneficiary of a social security scheme;
  * Subject falling into several categories above;
* Subject who refused to participate in the study;
* Subject participating in an interventional clinical study;
* Subject who, according to the investigator, has cognitive problems that prevent him/her from completing a questionnaire or for whom the assessment may be a problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Self-Questionnaire responses on final criteria for Coloplast catheter selection associated with patient satisfaction. | At 6 months.
  The primary objective of this study is to specify the final criteria for choosing the Coloplast catheter that provides patient satisfaction, as determined by self-questionnaire. Responses are scored ranging from 0 (strongly disagree) to 4 (strongly agree). Higher scores indicate a more positive attitude toward urinary self-catheterization.

SECONDARY OUTCOMES:
Self-Questionnaire responses on criteria for patient's initial Coloplast catheter selection choice. | Day 0 (at inclusion visit).
  Responses are assessed using the self-questionnaire, which evaluates the importance of various factors influencing catheter choice (e.g., comfort, packaging, ease of use, hygiene). Items are rated on a 4-point scale from 1 = Not at all important to 4 = Very important, with higher scores indicating greater importance assigned to that factor.
Five-Point scale scores for patient's satisfaction with Coloplast catheter. | At 3 to 12 weeks AND at 6 months.
  Satisfaction and ease of learning are each rated on 5-point scales, where higher scores denote higher satisfaction or greater ease.
Intermittent Catheterization Difficulty Questionnaire (IC-Di-Q) questionnaire scores for challenges in Intermittent Self-Catheterization (ISC). | At 3 to 12 weeks AND at 6 months.
  Responses are assessed with the Intermittent Catheterization Difficulty Questionnaire (IC-Di-Q), which evaluates the frequency and intensity of difficulties experienced during urinary self-catheterization over the past 15 days. Each item is rated on two 4-point scales: frequency (1 = Never to 4 = Always) and intensity (1 = None to 4 = Considerable). Higher scores indicate more frequent and/or more severe catheterization difficulties.
Patient's final choice criteria for the catheter selection variables. | At 6 months.
  Participants report the type of catheter most frequently used.
Adherence rates to Intermittent Self-Catheterization (ISC) protocol. | At 6 months.
  Participants report their average daily catheterization frequency compared to the prescribed regimen; higher self-reported adherence indicates better compliance with the ISC protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Houben, PhD MBA, Study Director — Coloplast A/S
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Background] Averbeck MA, Kennelly M, Thiruchelvam N, Konstantinidis C, Chartier-Kastler E, Krassioukov A, Landauro M, Jacobsen L, Vaabengaard R, Islamoska S. Risk factors for urinary tract infections associated with lower quality of life among intermittent catheter users. Br J Nurs. 2023 Oct 12;32(18):S8-S16. doi: 10.12968/bjon.2023.32.18.S8. PMID 37830866
- [Background] Kennelly M, Thiruchelvam N, Averbeck MA, Konstatinidis C, Chartier-Kastler E, Trojgaard P, Vaabengaard R, Krassioukov A, Jakobsen BP. Adult Neurogenic Lower Urinary Tract Dysfunction and Intermittent Catheterisation in a Community Setting: Risk Factors Model for Urinary Tract Infections. Adv Urol. 2019 Apr 2;2019:2757862. doi: 10.1155/2019/2757862. eCollection 2019. PMID 31065264
- [Background] Guinet-Lacoste A, Kerdraon J, Rousseau A, Gallien P, Previnaire JG, Perrouin-Verbe B, Amarenco G. Intermittent catheterization acceptance test (I-CAT): A tool to evaluate the global acceptance to practice clean intermittent self-catheterization. Neurourol Urodyn. 2017 Sep;36(7):1846-1854. doi: 10.1002/nau.23195. Epub 2017 Jan 16. PMID 28090660
- [Background] Chartier-Kastler E, Amarenco G, Lindbo L, Soljanik I, Andersen HL, Bagi P, Gjodsbol K, Domurath B. A prospective, randomized, crossover, multicenter study comparing quality of life using compact versus standard catheters for intermittent self-catheterization. J Urol. 2013 Sep;190(3):942-7. doi: 10.1016/j.juro.2013.04.026. Epub 2013 Apr 12. PMID 23587630
- [Background] Game X, Phe V, Castel-Lacanal E, Forin V, de Seze M, Lam O, Chartier-Kastler E, Keppenne V, Corcos J, Denys P, Caremel R, Loche CM, Scheiber-Nogueira MC, Karsenty G, Even A. Intermittent catheterization: Clinical practice guidelines from Association Francaise d'Urologie (AFU), Groupe de Neuro-urologie de Langue Francaise (GENULF), Societe Francaise de Medecine Physique et de Readaptation (SOFMER) and Societe Interdisciplinaire Francophone d'UroDynamique et de Pelvi-Perineologie (SIFUD-PP). Prog Urol. 2020 Apr;30(5):232-251. doi: 10.1016/j.purol.2020.02.009. Epub 2020 Mar 24. PMID 32220571
- [Background] Stensballe J, Looms D, Nielsen PN, Tvede M. Hydrophilic-coated catheters for intermittent catheterisation reduce urethral micro trauma: a prospective, randomised, participant-blinded, crossover study of three different types of catheters. Eur Urol. 2005 Dec;48(6):978-83. doi: 10.1016/j.eururo.2005.07.009. Epub 2005 Aug 2. PMID 16126331
- [Background] Salomon J, Gory A, Bernard L, Ruffion A, Denys P, Chartier-Kastler E. [Urinary tract infection and neurogenic bladder]. Prog Urol. 2007 May;17(3):448-53. doi: 10.1016/s1166-7087(07)92346-5. French. PMID 17622075
- [Background] Scotland KB, Lange D. Prevention and management of urosepsis triggered by ureteroscopy. Res Rep Urol. 2018 Jul 5;10:43-49. doi: 10.2147/RRU.S128071. eCollection 2018. PMID 30013956
- [Background] Herve F, Ragolle I, Amarenco G, Viaene A, Guinet-Lacoste A, Bonniaud V, Everaert K. Assessment of Intermittent Self-Catheterization Procedures in Patients with Neurogenic Lower Urinary Tract Dysfunction: Dutch Translation and Validation of the Intermittent Catheterization Satisfaction Questionnaire, Intermittent Catheterization Acceptance Test, Intermittent Self Catheterization Questionnaire and Intermittent Catheterization Difficulty Questionnaire. Urol Int. 2019;102(4):476-481. doi: 10.1159/000499884. Epub 2019 Apr 18. PMID 30999304
- [Background] Guinet-Lacoste A, Jousse M, Tan E, Caillebot M, Le Breton F, Amarenco G. Intermittent catheterization difficulty questionnaire (ICDQ): A new tool for the evaluation of patient difficulties with clean intermittent self-catheterization. Neurourol Urodyn. 2016 Jan;35(1):85-9. doi: 10.1002/nau.22686. Epub 2014 Oct 18. PMID 25327888
- [Background] Girotti ME, MacCornick S, Perisse H, Batezini NS, Almeida FG. Determining the variables associated to clean intermittent self-catheterization adherence rate: one-year follow-up study. Int Braz J Urol. 2011 Nov-Dec;37(6):766-72. doi: 10.1590/s1677-55382011000600013. PMID 22233982
- [Background] Thiruchelvam N, Hashim H, Forman CR, Jacobsen L, Sperup T, Andersen K. New compact micro-hole zone catheter enables women to achieve effective bladder emptying without flow-stops. Br J Nurs. 2024 Sep 19;33(17):834-843. doi: 10.12968/bjon.2024.0212. PMID 39302905
- [Background] Gabbe BJ, Nunn A. Profile and costs of secondary conditions resulting in emergency department presentations and readmission to hospital following traumatic spinal cord injury. Injury. 2016 Aug;47(8):1847-55. doi: 10.1016/j.injury.2016.06.012. Epub 2016 Jun 7. PMID 27343134
- [Background] Biering-Sorensen F. Urinary tract infection in individuals with spinal cord lesion. Curr Opin Urol. 2002 Jan;12(1):45-9. doi: 10.1097/00042307-200201000-00009. PMID 11753133
- [Background] Biering-Sorensen F, Bagi P, Hoiby N. Urinary tract infections in patients with spinal cord lesions: treatment and prevention. Drugs. 2001;61(9):1275-87. doi: 10.2165/00003495-200161090-00004. PMID 11511022
- [Background] Flores-Mireles AL, Walker JN, Caparon M, Hultgren SJ. Urinary tract infections: epidemiology, mechanisms of infection and treatment options. Nat Rev Microbiol. 2015 May;13(5):269-84. doi: 10.1038/nrmicro3432. Epub 2015 Apr 8. PMID 25853778
- [Background] Pascoe G, Clovis S. Evaluation of two coated catheters in intermittent self-catheterization. Br J Nurs. 2001 Mar 8-21;10(5):325-9. doi: 10.12968/bjon.2001.10.5.5360. PMID 12170675
- [Background] Chartier-Kastler E, Denys P. Intermittent catheterization with hydrophilic catheters as a treatment of chronic neurogenic urinary retention. Neurourol Urodyn. 2011 Jan;30(1):21-31. doi: 10.1002/nau.20929. Epub 2010 Oct 6. PMID 20928913